CLINICAL TRIAL: NCT02113995
Title: Clinical Evaluation, Organic Response in Obesity Patients Subjected to Vertical Videolaparoscopy Gastroplasty With or Without Perioperative Cares Recommended by the Acerto Project.
Brief Title: Clinical Evaluation, Organic Response in Obesity Patients Subjected to Vertical Videolaparoscopy Gastroplasty With or Without Perioperative Cares Recommended by the Acerto Project. Randomized Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cuiaba University (Other)
Responsible Party: Principal Investigator, Gunther Peres Pimenta, MD PhD Gunther Peres Pimenta, Cuiaba University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 018/CEP-UNIC/2011.
Record Dates: First submitted 2014-04-12; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: To Evaluate Clinical Results, Insulin Resistance and Inflammatory Response to Trauma in Morbidly Obese Patients
Keywords: Obesity, Morbid; Insulin Resistance; Acute-Phase Reaction; Gastroplasty; Length of Stay; Protocols; Randomized Controlled Trial.
MeSH Terms: conditions — Insulin Resistance; Obesity, Morbid; Acute-Phase Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACERTO (Active Comparator): Patients received 400 ml of a beverage containing water and 50 g of maltodextrin 6 hours before the operation. They received orally extra 200 ml of this beverage containing water and 25 g of maltodextrin 3 hours before the operation. Regarding the intravenous fluids, they received 1 to 1.5 liter of crystalloid fluids (ringer lactate) in the intraoperative. In the immediate postoperative they were programmed to receive 2 liters of crystalloid fluids (ringer lactate) and 1 to 2 liters in the first day of the postoperative period. The venous hydration was suspended as soon as they started to drink liquids.
  Prophylaxis of nausea and vomiting with dexamethasone 8 mg at the beginning of the anesthesia and ondansetron 4-8 mg after the surgery. In the postoperative period we utilized analgesics such as dipyrone and ketorolac and, if necessary, low doses of morphine and antiemetics like ondansetron.
  Interventions: Other: ACERTO protocol vs Traditional care
- Traditional care (Active Comparator): The analgesia in the postoperative period of the group control was performed with dipyrone, tramadol hydrochloride, and morphine. The prophylaxis of nausea and vomiting with dexamethasone 8 mg in the beginning of the anesthesia and the metoclopramide at the end of the surgery. During the anesthetic induction antibiotic prophylaxis (cefazolin 3 grams/day for 2 days) was administrated.
  The control group were submitted to the protocol of traditional fasting with at least 8 hours. Patients in this group received 1 to 2 liters of crystalloid fluid (ringer lactate) in the intraoperative, and they received 3 to 4 liters of crystalloid fluids (ringer lactate, saline 0.9% and/or dextrose 5%). In the immediate postoperative, 2 to 3 liters in the first day of postoperative and, finally, 1 to 2 liters in the second day of the postoperative.
  Interventions: Other: ACERTO protocol vs Traditional care

INTERVENTIONS:
Other: ACERTO protocol vs Traditional care — Three sample blood collections were performed, being one in the anesthesic induction and the others in the next 24 to 48 hours. The blood was sent to the laboratory for dosages of glucose, insulin, C-reactive protein, albumin, prealbumin, alpha 1 acid glycoprotein and interleukin 6. During the anesthesic induction we also collected blood for analize glycosylated hemoglobin.

SUMMARY:
Background To evaluate clinical results, insulin resistance and inflammatory response to trauma in morbidly obese patients undergoing laparoscopic Sleeve gastrectomy who received either traditional preoperative care or treatment following the ACERTO protocol.

DETAILED DESCRIPTION:
Methods The population of the study consisted of morbidly obese patients, who were operated on with the Sleeve procedure, from Cuiaba, MT, between April and October 2012. We studied the inflammatory response and insulin resistance by measuring levels of glucose, insulin, Homa IR, reactive C protein, albumin, pre-albumin, alpha 1 acid glicoprotein, interleukin 6 and glycosylated hemoglobin. We also studied hydration, nausea and vomiting, hypertension, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria: We included patients who are between 18 and 45 years of age, from both sexes, with an initial BMI (Body Mass Index) which is equal to or greater than 40 kg/m2, candidates for the sleeve surgery procedure through laparoscopy.

-

Exclusion Criteria: We excluded the patients who didn't follow the fasting protocol and also those whose laboratory exams were lost.

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
ACERTO protocol | 6 months
  To evaluate clinical results, insulin resistance and inflammatory response to trauma in morbidly obese patients undergoing laparoscopic Sleeve gastrectomy who received either traditional preoperative care or treatment following the ACERTO protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Gunther P Pimenta, MD, PhD, Principal Investigator — Cuiaba University
Locations (1):
- ACERTO protocol, Cuiabá, Mato Grosso, Brazil